CLINICAL TRIAL: NCT05591573
Title: The Impact of Glycemic Index on Sleep and Memory Consolidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Dr Hayley Young, Associate Professor, Swansea University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SSSU
Record Dates: First submitted 2022-07-15; First posted 2022-10-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Sleep Architecture; Cognitive Function; Mood; Glucose Metabolism

STUDY DESIGN:
Intervention Model Description: In a randomized, double-blind, and counterbalanced order (AB/BA), participants will receive either a high glycemic index or low glycemic index pre-bed drink. After a 1-week washout period, participants will consume the alternate drink.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To ensure blinding of participants and researchers, a randomisation list will be produced using Statistical Package for the Social Sciences (SPSS) software by an employee of Swansea University, who is not actively involved in the study.
  Blinding will be maintained by the use of encoded beverages to ensure participants, researchers, and the data analysers are unaware of the intervention. The blind will be broken only after statistical analysis of the data is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low glycemic index drink (Experimental): Fruit drink containing low glycemic index sugar.
  Interventions: Dietary Supplement: Low glycemic index drink
- High glycemic index drink (Experimental): Fruit drink containing high glycemic index sugar.
  Interventions: Dietary Supplement: High glycemic index drink

INTERVENTIONS:
Dietary Supplement: Low glycemic index drink — Fruit flavoured drink with low glycemic index sugar (300 ml)
  Arms: Low glycemic index drink
Dietary Supplement: High glycemic index drink — Fruit flavoured drink with high glycemic index sugar (300 ml)
  Arms: High glycemic index drink

SUMMARY:
The study will test whether the consumption of a low versus a high glycemic index pre-bed drink influences sleep architecture, memory consolidation, nocturnal glucose metabolism, and mood.

DETAILED DESCRIPTION:
Few studies have examined the impact of meal composition on sleep. Most research has focused on carbohydrate intake, although reports are sporadic and confounded by the manipulation of other macronutrients. Nonetheless, the pattern of results appears to depend on the nature of the sleep variable under investigation e.g., latency, duration, or efficiency. The study will determine whether manipulating the glycemic index of a pre-bed drink influences sleep architecture, procedural and declarative memory consolidation, nocturnal glucose metabolism, and mood.

Participants will stay in the sleep laboratory for three nights, each night separated by one week (visit 1, 2, and 3). The first night is an acclimatisation night. The same procedure will be followed on all three nights, as described below.

On the morning of each visit, a continuous glucose monitor will be set up and worn until 8pm the following evening. Participants will be asked to return to the sleep laboratory at 7pm, having fasted for five hours, and asked to consume a standardised evening meal. Several mood questionnaires will be completed throughout the evening and a polysomnography will be set up. Two memory tasks will be administered at approximately 10pm. Immediately after this, participants will consume either water (night 1), or a low glycemic index or high glycemic index drink (night 2 or 3). Participants will retire to bed at approximately 11pm and woken up between 6.30am - 8am, depending on personal preference.

In the morning, the memory tasks will be administered again, as well as two mood questionnaires. Participants will be asked to wear a Pro-Diary watch throughout the day, which measures mood and hunger. At 8pm, both the continuous glucose monitor and Pro-diary watch will be collected from the participant.

ELIGIBILITY:
Inclusion Criteria:

* Male (given that the menstrual cycle may influence sleep polysomnography)
* Good health
* Not taking any medication known to effect sleep or metabolism
* Normal sleep duration (i.e. between 6.5 - 9 hours of sleep per night)
* A sleep efficiency score above 80% (Pittsburg Sleep Quality Index)
* Normal sleep schedule (i.e. fall asleep between 10pm and 12pm)
* No difficulty sleeping in new places

Exclusion Criteria:

* Diagnosis of any physical or mental disorder e.g. diabetes, cardiovascular disorders, gastrointestinal disorders, sleep problems, epilepsy, or mood disorders
* Unhealthy weight (BMI over 30)
* Drink more than 300mg of caffeine per day (3 - 4 standard sized 8-oz cups)
* Work nights or shifts
* Smoke/vape
* Regularly drink alcohol (>3 glasses per day)
* Used recreational drugs within the last 6 months
* Take part in >3 hours of vigorous exercise per week
* Any known food allergies or intolerances
* Nocturnal eating or regular consumption of alcohol before bed (assessed by the Meal Pattern Questionnaire)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-31 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Sleep onset latency (polysomnography) | Bedtime (approx. 11.00pm) to wake time (approx 7.30am)
  Onset of sleep from the time the lights are turned off.
Total sleep time (polysomnography) | Bedtime (approx. 11.00pm) to wake time (approx 7.30am)
  The total number of hours of sleep.
Wake after sleep onset (polysomnography) | Bedtime (approx. 11.00pm) to wake time (approx 7.30am)
  Hours of wake time after three epochs of sleep have occurred.
Sleep efficiency (polysomnography) | Bedtime (approx. 11.00pm) to wake time (approx 7.30am)
  Total sleep time divided by the time from lights out until awakening in the morning.
Sleep stages (polysomnography) | Bedtime (approx. 11.00pm) to wake time (approx 7.30am)
  Time spent in each sleep stage.
Arousal index (polysomnography) | Bedtime (approx. 11.00pm) to wake time (approx 7.30am)
  Number of arousals throughout the night.
Leeds Sleep Evaluation Questionnaire | Administered 10 - 20 minutes after waking up in the morning,
  Subjective assessment of sleep quality. Scores range from 0 to 30. Higher scores indicate poorer sleep quality.

SECONDARY OUTCOMES:
Glucose response (continuous glucose monitor) | 25 hours during night 2 and night 3 (weeks 2 and 3)
  The 2h and 3h incremental area under the curve (iAUC) will be used to assess glycemic response to the pre-bed drink. The mean amplitude of glycemic excursion (MAGE) will be assessed as an indicator for glycemic variability during the night and for 25 hours.
Finger tapping task (procedural memory) | Completed at 10pm, and between 6.30 - 8am the following morning, on night 2 and night 3 (week 2 and 3).
  The change in performance from the learning phase to the recall phase.
Story recall task (declarative memory) | Completed at 10pm, and between 6.30 - 8am the following morning, on night 2 and night 3 (week 2 and 3).
  The number of content words (nouns, adjectives, and verbs) correctly recalled.
Epworth Sleepiness Scale | Administered at 8pm on the evening after night 2 and night 3 (week 2 and 3).
  Subjective assessment of daytime sleepiness. Scores range from 0 - 24. Higher scores indicate more daytime sleepiness.
Mood and hunger | Completed five times throughout the evening and twice in the morning (immediately after waking up and 20-30 minutes later) on night 2 and night 3 (week 2 and 3). .
  Scores range from 0 - 100. Higher scores indicate stronger feelings.
Mood | Prompted from 9.30am - 5.30pm after night 2 and night 3 (week 2 and 3).
  Pro-diary watch
Actigraphy | Night 2 and night 3 (week 2 and 3).
  Time spent in each sleep stage.

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Young, Study Director — Swansea University
Locations (1):
- Swansea University, Swansea, West Glamorgan, United Kingdom

REFERENCES:
- [Derived] Gaylor CM, Brennan A, Blagrove M, Tulip C, Bloxham A, Williams S, Tucker R, Benton D, Young HA. Low and high glycemic index drinks differentially affect sleep polysomnography and memory consolidation: A randomized controlled trial. Nutr Res. 2025 Feb;134:49-59. doi: 10.1016/j.nutres.2024.11.012. Epub 2024 Dec 4. PMID 39854800